CLINICAL TRIAL: NCT07245498
Title: Efficacy of Extracorporeal Shock Wave Therapy in Chronic Non-radicular Low Back Pain
Brief Title: ESWT for Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TABED 2-24-246
Record Dates: First submitted 2025-10-01; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain; Physical Therapy; Extracorporeal Shock Wave Therapy
Keywords: low back pain,; Extracorporeal shock wave therapy; Conventional physical therapy
MeSH Terms: conditions — Low Back Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Group 1: Radial ESWT+conventional physical therapy+exercise Group 2: sham ESWT+conventional physical therapy+exercise Assesments: before treatment, after treatment and 1th month after treatment primer outcome: VAS seconder outcomes: Oswestry disability index, hospital axiety and depression scale
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ekstra corporeal shock wave therapy(ESWT) (Active Comparator): Ekstra corporeal shock wave therapy + conventional physical therapy +exercise
  Interventions: Other: extracorporeal shock wave therapy
- sham Ekstra corporeal shock wave therapy (Sham Comparator): sham Ekstra corporeal shock wave therapy+ conventional physical therapy +exercise
  Interventions: Other: extracorporeal shock wave therapy

INTERVENTIONS:
Other: extracorporeal shock wave therapy — Shock wave probe applied perpendicularly to the quadratus lumborum, the sacroiliac joint, and the regions of the patient's lumbar area where pain is localized, following the application of coupling gel to facilitate the transmission of pressure waves generated by the device through the skin via its metallic applicator head

SUMMARY:
The goal of this interventional study is to compare the effects of ESWT in women and men between the age 18-65 with non radicular non specific low back pain . The main question it aims to answer is:

Is intervention ESWT more effective than conventional physical therapy agents. Patients were divided into 2 groups; Group 1 ESWT+conventional physical therapy and group 2: sham ESWT+conventional physical therapy. Study follow up time before treatment, 0 week after treatment, and 1 month after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 65 who have had low back pain for at least three months and have been diagnosed with chronic low back pain.
* Patients who consent to participate in the study according to the informed consent form will be included in the study.

Exclusion Criteria:

* Diagnosis of spondylolisthesis, spondylolysis, spinal tumors, intervertebral disc infections, severe osteoporosis, or lumbar vertebral fractures and patients with a history of prior spine surgery,
* Currently using anti-inflammatory drugs or analgesics in last four weeks,
* Local skin infection or damage at the treatment site,
* Inflammatory rheumatic diseases,
* Pregnancy
* Concomitant mental diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale(VAS) | Before treatment, Baseline and 1month after treatment
  The VAS is a validated tool for assessing pain intensity. It consists of a 10-cm horizontal line anchored by "no pain" (0) at the left end and "worst imaginable pain" (10) at the right end. Participants indicate their perceived pain level by marking a point on the line, which is then measured in centimeters to provide a continuous pain score from 0 to 10.

SECONDARY OUTCOMES:
oswestry disability score(ODI), | Before treatment, Baseline, 1st month after treatment
  The ODI is a widely used, validated questionnaire designed to measure disability related to low back pain. It consists of 10 sections covering domains such as pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and employment/homemaking. Each section is scored from 0 to 5, with higher scores indicating greater disability. The total score is expressed as a percentage, with 0% representing no disability and 100% representing maximum disability.
hospital anxiety and depression scale(HADS) | Before treatment, Baseline, 1st month after treatment
  The HADS is a self-administered questionnaire developed to detect states of anxiety and depression in patients with physical health problems. It consists of 14 items, divided into two subscales: anxiety (HADS-A, 7 items) and depression (HADS-D, 7 items). Each item is scored on a 4-point scale (0-3), giving a maximum score of 21 for each subscale. Higher scores indicate greater levels of anxiety or depression, with established cutoffs used to classify symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Çankaya, Turkey (Türkiye)